CLINICAL TRIAL: NCT00920322
Title: A Randomised Study of rTMS in Depression
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Technical issues impeded recruitment.
Sponsor: Northside Clinic, Australia (Other)
Responsible Party: Associate Professor Colleen Loo, University of NSW
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSG HREC 153; UNSW HREC 9074
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Depression
Keywords: Depression; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- five times weekly (Active Comparator): Patients will receive rTMS on each weekday for 4 weeks (5 x weekly)
  Interventions: Device: rTMS 5 x weekly
- three times weekly (Experimental): Patients will receive rTMS three times weekly for four weeks
  Interventions: Device: rTMS 3 times weekly

INTERVENTIONS:
Device: rTMS 5 x weekly — Patients will receive rTMS five times weekly for 4 weeks
  Arms: five times weekly
Device: rTMS 3 times weekly — Patients will receive rTMS 3 times weekly for 4 weeks
  Arms: three times weekly

SUMMARY:
This study will report on the outcomes of rTMS administered 3 times per week, compared with the standard protocol of 5 times per week. Participants will be randomly assigned to frequency condition and depressive symptomatology will be measured weekly using a range of clinician and self-rated questionnaires. Participants will remain in the study for at least 4 weeks, with the option of continuing for a further 2 weeks as judged by the study psychiatrist. It is hypothesised that rTMS administered three times per week will be equally as effective as rTMS administered five times per week in reducing depressive symptomatology.

DETAILED DESCRIPTION:
Numerous studies have demonstrated the efficacy of active rTMS over sham rTMS for depression; however, few have systematically studied the optimal frequency of treatment sessions to achieve this efficacy. To date, the majority of studies have administered rTMS every weekday, although this approach has not been widely contested. In addition, most studies have only assessed the effectiveness of rTMS over a two week period, which has resulted in some improvement in depressive symptomatology; however, a longer treatment course would likely result in greater improvement. In this study depressed patients will be randomly assigned to receive rTMS either 3 or 5 times per week, for a period of 4-6 weeks. A range of rating scales will be used to assess the improvement of depressive symptomatology within and between the two frequency groups, to ultimately determine whether TMS is needed 5 times per week to achieve adequate anti-depressant effects or whether 3 times per week is sufficient in achieving a similar level of efficacy for patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged >/= 18
* DSM-IV diagnosis of Major Depressive Episode (bipolar or MDD)
* MADRS score >/= 20
* Able to give informed consent
* Psychoactive medication dosages have been stable for a period of 4 weeks prior to entry in the study

Exclusion Criteria:

* Co-morbid alcohol or drug abuse or dependence (last 3 months), current eating disorder, mental retardation, schizophrenia, rapid cycling bipolar
* A history of mood 'switching' in response to other treatments, which cannot be contained by concurrent treatment, e.g., mood stabiliser
* Pregnancy
* Significant neurological disorder that increases seizure risk
* Metal objects in the head, pacemakers, or a history of epilepsy
* Patients who have failed to respond to a course of ECT in their current episode of depression
* A high risk of suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Depression Rating Scales | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, MBBS, FRANZCP, MD, Principal Investigator — University of NSW
Locations (1):
- Northside Clinic, Greenwich, New South Wales, Australia